CLINICAL TRIAL: NCT03686046
Title: Evaluation of an Open-source Speech-processing Platform
Acronym: EOSP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Diego State University (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Arthur Boothroyd, Professor, San Diego State University
Other Study IDs: 58786
Record Dates: First submitted 2018-08-02; First posted 2018-09-26 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Hearing aid
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exploratory use: Brief (2 hour) exploratory use of prototype self-adjusted wearable Master Hearing Aid
  Interventions: Other: Exploratory use

INTERVENTIONS:
Other: Exploratory use — Participants will be accompanied by a researcher while wearing the open-source speech processing platform as a hearing aid - adjusted to their needs using a widely accepted Fitting prescription. Using a hand-held controller, they will readjust to their liking as the acoustic conditions change. After returning to the laboratory, they will complete speech perception tests using under their self-selected amplification conditions and respond to a structured interview dealing with perceived performance of the device and its acceptability as a hearing aid during possible field studies.

SUMMARY:
Determining acceptability and usability of a wearable open-source speech processing platform (Master Hearing Aid) developed for hearing-aid research

DETAILED DESCRIPTION:
Part 1 Speech perception tests. You will hear words and sentences under a variety of listening conditions and be asked either to either repeat them or to select what you heard from a set of options. You will also answer a few questions about the speech and the background noise. The goal is to determine the ability of the most recent version of the device to deliver good quality speech that is comfortable and understandable over a range of conditions that are representative of everyday listening.

Part 2. Suitability and Acceptability. You will be asked to respond to a short structured interview about the device. If the device has reached a wearable stage, you will wear it outside the laboratory while engaging in discussion with one of the researchers before completing the interview. The goal is to obtain the opinions of persons with hearing loss about the device itself, and about their willingness to wear it as a hearing aid in their everyday life, if they were to be involved in a research study.

Part 3 is a focus-group session with about 10 hearing-aid users, some of whom will have participated in Parts 1 and 2. Topics will deal with hearing aids in general and about the current version of the experimental device. Discussion will be recorded for later transcription and analysis. The goal is to gain the perspective of hearing-aid users about hearing aids, hearing-aid research, and the acceptability of this experimental device for field research.

ELIGIBILITY:
Inclusion Criteria:

- Sensorineural hearing loss

Exclusion Criteria:

* Cognitively challenged
* Legally blind

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with sensorineural hearing loss Residents of San Diego county and North county, California
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Response to structured interview | Approximately 2 weeks after last participant completes the exploratory use, estimated to be about 6 months.
  A wearable speech-processing platform for hearing-aid research
  1. How long might you be prepared to wear this device as a hearing aid for purposes of research?
  2. How do you rate the appearance and wearability of the device?
  3. How do you rate the performance of the device as a hearing aid?
  4. What changes might increase your willingness to wear this device for research purposes?
  5. What changes might increase your rating of appearance?
  6. What changes might increase your rating of performance?

SECONDARY OUTCOMES:
Electro-acoustic performance of the speech-processing platform | Approximately 2 weeks after last participant completes the exploratory use, estimated to be about 6 months.
  Real-ear gain versus frequency curves of the speech-processing platform, before and after self-adjustment during the brief trial, will be obtained with the Verifit 2 hearing-aid test system - using standard audiological clinical procedures. (Mackersie, Boothroyd and Lithgow, 2018).
Aided speech perception | Approximately 2 weeks after last participant completes the exploratory use, estimated to be about 6 months.
  Participants will repeat prerecorded single syllable words presented at varying levels levels from a loudspeaker. Performance will be assessed as the percentage of speech sounds correctly repeated and will be measured while wearing the speech-processing platform as set before and after self-adjustment. (Boothroyd, 2008)
Pattern of user self-adjustments. | Approximately 2 weeks after last participant completes the exploratory use
  Changes of gain and spectral slope initiated by participants in response to changing , estimated to be about 6 months.acoustic conditions will be automatically logged by the self-adjustment software. (Boothroyd and Mackersie (2017)
Participant-specified issues, comments, and opinions | Approximately 2 months after last participant completes the exploratory use, estimated to be about 6 months.
  Focus group for all participants

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Boothroyd, Ph.D, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, Audiology Clinic, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boothroyd A, Mackersie C. A "Goldilocks" Approach to Hearing-Aid Self-Fitting: User Interactions. Am J Audiol. 2017 Oct 12;26(3S):430-435. doi: 10.1044/2017_AJA-16-0125. PMID 29049625
- [Result] Mackersie C, Boothroyd A, Lithgow A. A "Goldilocks" Approach to Hearing Aid Self-Fitting: Ear-Canal Output and Speech Intelligibility Index. Ear Hear. 2019 Jan/Feb;40(1):107-115. doi: 10.1097/AUD.0000000000000617. PMID 29894379
- [Result] Lee CH, Kates JM, Rao BD, Garudadri H. Speech quality and stable gain trade-offs in adaptive feedback cancellation for hearing aids. J Acoust Soc Am. 2017 Oct;142(4):EL388. doi: 10.1121/1.5007278. PMID 29092590
- [Result] Boothroyd A. The performance/intensity function: an underused resource. Ear Hear. 2008 Aug;29(4):479-91. doi: 10.1097/AUD.0b013e318174f067. PMID 18469711